CLINICAL TRIAL: NCT05781373
Title: Effect of Intraoperative PEEP Individualization According to Driving Pressure in Major Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor head of anesthesia and intensive care department, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: individualized Peep
Record Dates: First submitted 2023-03-01; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed PEEP group (No Intervention): Protective intraoperative ventilation with: 6 ml/kg IBW tidal volume recruitment maneuver and fixed PEEP¨level of 6 cmH2O
- Individualized PEEP group (Experimental): Protective intraoperative ventilation with: 6 ml/kg IBW tidal volume recruitment maneuver and individualized PEEP¨level in order to achieve the lowest driving pressure
  Interventions: Procedure: Peep individualization

INTERVENTIONS:
Procedure: Peep individualization — Intraoperative Peep individualization in order to achieve the lowest driving pressure
  Arms: Individualized PEEP group

SUMMARY:
In this prospective, randomized trial, including patients scheduled for a major open or laparoscopic abdominal surgery (duration >2 hours) under general anesthesia , the investigators will compare 2 strategies of protective mechanical ventilation: a fixed intraoperative PEEP of 6 cmH2O and an individualized intraoperative PEEP according to the driving pressure.

DETAILED DESCRIPTION:
Patients will be randomized into 2 groups:

* Fixed PEEP group: will receive protective intraoperative mechanical ventilation: tidal volume: 6 ml/kg of PBW, recruitment maneuvers every immediately after tracheal intubation and every 2 hours and a fixed PEEP of 6 cmH2O
* Individualized PEEP: protective mechanical ventilation with the same modality with an individualization of PEEP levels hourly in order to achieve the lowest driving pressure. PEEP levels will be adjusted after intubation and hourly by increasing or decreasing PEEP levels every 10 respiratory cycles.

The primary outcome: incidence of post operative pulmonary complications during the first post operative days.

ELIGIBILITY:
Inclusion Criteria:

* BMI<35, ARISCAT score > 26, patients scheduled for major abdominal surgery

Exclusion Criteria:

* unplanned post operative ICU stay and mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
incidence of pulmonary post operative complications | first 7 post operative days
  SpO2< 92%, new chest Xray infiltrates, acute respiratory failure requiring intervention

SECONDARY OUTCOMES:
lung aeration score (LAS) | day 1, day 3 and day 7 after surgery
  assessment LAS with lung ultrasound minimum 0 maximum: 36 (worse outcome)

IPD SHARING:
Plan to Share IPD: No